CLINICAL TRIAL: NCT06312735
Title: Cluster-randomized Controlled Trial of Virtual Reality for Patients With Chronic Musculoskeletal Pain (Wait & Work)
Brief Title: VR for Patients With Chronic Pain (Wait & Work)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Monique Tabak, Professor, University of Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 230405
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Four-week, at-home VR intervention with a recommended daily use of 10-30 minutes
  Interventions: Device: VR (Reducept)
- Control group (No Intervention): No intervention, patient is a waiting-list control

INTERVENTIONS:
Device: VR (Reducept) — Reducept is a novel VR intervention that consists of a combination of pain neuroscience education (PNE) and pain management techniques. It includes different psychological therapy modalities (e.g. acceptance and commitment therapy (ACT), cognitive behavioral therapy (CBT) and hypnotherapy) into a single application.
  Arms: Intervention group

SUMMARY:
This cluster-RCT evaluates the effect of therapeutic virtual reality (VR) on patients with chronic musculoskeletal pain (CMP) who are on a waiting list to receive pain treatment. The used VR application, Reducept, offers pain education and pain management techniques. This home-based, stand-alone, immersive VR intervention was used daily for four weeks in the intervention group. The control group received standard care (no treatment). Primary outcome measure for this study was health-related quality of life, secondary outcome measures included various pain-related variables (e.g. pain self-efficacy and acceptance. Outcome variables will be measured after four weeks and follow-up after six months.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* suffering from primary or secondary CMP
* finished with biomedical diagnostics and treatment
* open to biopsychosocial treatment
* willing and capable of complying with study procedures.

Exclusion Criteria:

* not able to finish the VR intervention due to physical (e.g. visual impairment), mental (e.g. severe sensitivity to stimuli) or practical problems (e.g. insufficient tech-literacy)
* unable to finish Dutch questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in quality of life measured using the short-form 12 (SF-12) | Baseline, directly after the intervention, and at six months follow-up
  This questionnaire on quality of life scores from 12 (worst possible score) to 56 (best possible score)

SECONDARY OUTCOMES:
Change in pain intensity measured using the numeric pain rating scale (NPRS) | Baseline, directly after the intervention, and at six months follow-up
  This questionnaire on pain intensity scores from 0 (best possible score) to 100 (worst possible score)
Change in pain catastrophizing measured using the pain catastrophizing scale (PCS) | Baseline, directly after the intervention, and at six months follow-up
  This questionnaire on pain catastrophizing scores from 0 (best possible score) to 52 (worst possible score).
Change in pain self-efficacy measured using the pain self-efficacy questionnaire (PSEQ) | Baseline, directly after the intervention, and at six months follow-up
  This questionnaire scores from 0 (worst possible score) to 60 (best possible score).
Change in pain acceptance measured using the chronic pain acceptance questionnaire (CPAQ-8) | Baseline, directly after the intervention, and at six months follow-up
  This questionnaire scores from 0 (worst possible score) to 48 (best possible score).
Change in feelings of anxiety and depression measured using the hospital anxiety and depression scale (HADS) | Baseline, directly after the intervention, and at six months follow-up
  This questionnaire scores from 0 (worst possible score) to 42 (best possible score).
Change in quality of care measured using the client satisfaction questionnaire (CSQ-8) | Baseline, directly after the intervention, and at six months follow-up
  This questionnaire scores from 8 (worst possible score) to 32 (best possible score).
Change in medication use measured using an open-ended question | Baseline, directly after the intervention, and at six months follow-up
  This question inquires about current medication use

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Roessingh rehabilitation center, Enschede, Overijssel
  - Nocepta, Hengelo, Overijssel
  - Revalidatie Friesland, Emmeloord, Provincie Friesland

IPD SHARING:
Plan to Share IPD: No